CLINICAL TRIAL: NCT02474706
Title: Evaluation of the Non-inferiority of Cefoxitin Versus Imipenem/Cilastatin in the Treatment of Urinary Tract Infections Caused by ESBL-producing Escherichia Coli
Acronym: COLIFOX
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC N 2013/COLIFOX-MAY/SR
Record Dates: First submitted 2015-06-04; First posted 2015-06-18 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Urinary Tract Infections
Keywords: cefoxitin Patient safety; Infectious diseases; Extended-Spectrum β-lactamases E.coli; Antibiotics
MeSH Terms: conditions — Urinary Tract Infections; Communicable Diseases | interventions — Cefoxitin; Imipenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cefoxitin (Experimental): Cefoxitin 2 g administered intravenously three times a day. during 10 days for the treatment of pyelonephritis during 21 days for the treatment of prostatitis
  Interventions: Drug: Cefoxitin
- imipenem (Active Comparator): Imimpenem 1 g administered intravenously three times a day. during 10 days for the treatment of pyelonephritis during 21 days for the treatment of prostatitis
  Interventions: Drug: imipenem

INTERVENTIONS:
Drug: Cefoxitin
  Arms: cefoxitin
Drug: imipenem
  Arms: imipenem

SUMMARY:
Background Information: Infections caused by extended-spectrum β-lactamase (ESBL)-producing Escherichia coli are becoming increasingly common owing to incorrect use of antibiotics and cross-transmission in healthcare establishments. These give rise to major problems in standard clinical practice: penicillins and cephalosporins cannot be used, and resistance to the other classes of antibiotics normally used, such as fluoroquinolones or cotrimoxazole, is very frequently observed. The current therapeutic strategy involves the use of a carbapenem, which represents the last effective solution on an individual level. However, the growing use thereof is contributing, collectively, to the development of resistance due to the production of carbapenemases, which will become a major public health problem, with a potential therapeutic dead-end. This observation is particularly worrying due to the very small number of antibiotic agents currently in development.

Infectious disease specialists and microbiologists are thus examining alternative agents to carbapenems in the management of infections caused by ESBL-producing E. coli. One of the avenues which could be developed is the use of known agents, already on the market, which are active in vitro on ESBL-producing E. coli, but which are not currently recommended for this indication in standard practice due to the lack of conclusive studies. Cefoxitin, an antibiotic belonging to the cephamycin group, could thus represent an alternative of particular interest in the treatment of infections caused by ESBL-producing E. coli, and help limit the use of carbapenems.

The implementation of a prospective, randomized, non-inferiority study on ertapenem and cefoxitin is of the most interest from a methodological perspective. It will enable recommendations to be drawn up, with a high level of evidence, very long-awaited in the field.

Primary objective: To evaluate the bacteriological non-inferiority of cefoxitin versus imipenem in the treatment of non-severe urinary tract infections (other than cystitis) caused by ESBL-producing E. coli susceptible in vitro to cefoxitin.

Secondary objectives:

* To evaluate the clinical non-inferiority of cefoxitin versus imipenem in the treatment of non-severe urinary tract infections (other than cystitis) caused by ESBL-producing E. coli susceptible in vitro to cefoxitin.
* To evaluate the impact of cefoxitin and imipenem on the emergence of multiresistant bacteria in the gut flora.

DETAILED DESCRIPTION:
Rationale:

Commensal enterobacteriaceae of the digestive tract, mostly represented by E.coli, can cause a wide range of infections such as urinary tract infections or severe bacteraemia. For several years now, the misuse of antibiotics and cross-transmission in hospitals have led to the emergence of Enterobacteriaceae producing extended-spectrum β-lactamases (ESBL). The rising prevalence of ESBL is estimated at 8.2% in healthcare settings and at 6.2% in the community.

Carbapenems are considered the reference treatment for ESBL-producing E.coli (EESBL) infections. They often remain the last effective treatment on an individual level. But on a larger scale, their increasing use contributes to the emergence of resistance that might soon become a major public health issue.

Although the prevalence of ESBL remains low, the rate of ESBL epidemics in French hospitals has increased hugely since 2004. This could become a cause of concern especially because very few antibacterial agents are currently in development.

So infectiologists and microbiologists have to consider alternatives to carbapenems to treat infections caused by EESBL, which is stipulated in the new recommendations from the French High Council for Public Health and the Infectious Disease Society of America.

Older and well-known molecules that have proved to be effective in-vitro against EESBL may be an option. However due to a lack of conclusive studies, they're still not recommended in these cases. Cefoxitin, a cephamycin antibiotic, may be a good alternative treatment for EESBL infections and contribute to spare the use of carbapenems.

Originality and innovation:

Previous studies of cephamycins have shown encouraging results, but they were mostly cohort trials with retrospective data or subsets of non-randomized studies. So a randomized prospective non-inferiority study comparing ertapenem and cefoxitine is necessary. If the results show non-inferiority of cefoxitine versus ertapenem, immediate clinical application should ensue and lead to new recommendations, highly anticipated by the infectiologists who support this project via their clinical research network.

Project feasibility:

The pace of inclusions has been calculated based on recent data on cefoxitine, trimethoprim/sulfamethoxazole and ciprofloxacin sensitivity EESBL, 68% of EESBL are susceptible to céfoxitine and resistant to trimethoprim/sulfamethoxazole and ciprofloxacin. In 2011, 16 French laboratories, involved in the EARSS network, isolated 582 EESBL strains from blood culture. In the university hospital of Nancy, 205 EESBL strains were isolated from urine cultures in 2012. The challenge of including 250 patients with ESBL E.coli positive urine culture, in 18 months and in about 20 participating French centers, seems highly feasible.

Recent data showed that 68% of EESBL are susceptible to céfoxitine and resistant to trimethoprim/sulfamethoxazole and ciprofloxacin. In the university hospital of Nancy, 205 EESBL strains were isolated from urine cultures in 2012. The challenge of including 250 patients with ESBL E.coli positive urine culture, in 18 months and in about 20 participating French centers, seems highly feasible.

Expected benefits for patients and/or public health Immediate benefits are expected, on an individual level and on a wider scale. Indeed for the patient, the use of narrow-specturm antibiotics, but with an equivalent efficacy, decreases the risk of selecting even more highly resistant bacteria than EESBL in the digestive tract, such as carbapenemase-producing enterobacteriaceae (CPE). A patient colonized with CPE is at high risk of developing a CPE infection and the rates of recovery are low because of the small number of antibiotics that remain effective.

At the community level, the main challenge is the preservation of carbapenems (one of the last families of antibiotics still effective in the treatment of ESBL infections), and the restriction of its usage to the treatment of severe infections only. The increasing use of carbapenems generates a high selection pressure on enterobacteriaceae which results in a worrying increase of the prevalence of CPE. Moreover, the few remaining effective antimicrobials induce high rates of side effects. The assessment of the non-inferiority of older, well-known and active molecules such as cefoxitin is a highly anticipated and encouraging research area, especially because the molecules currently under development are far from being on the market.

Title: Non-inferiority study of cefoxitin versus imipenem as treatment for non-severe urinal tract infections (excluding cystitis) caused by extended spectrum beta-lactamases producing E.Coli susceptible to cefoxitin in-vitro

Primary objective: to show the bacteriological non-inferiority of cefoxitin versus imipenem as a treatment for non-severe urinary tract infections (excluding cystitis) caused by extended spectrum beta-lactamases producing E.Coli susceptible to cefoxitin in-vitro

Secondary objectives:

* to show the clinical non-inferiority of cefoxitin versus imipenem as a treatment for non-severe urinary tract infections (excluding cystitis) caused by extended spectrum beta-lactamases producing E.Coli susceptible to cefoxitin in-vitro
* to evaluate the impact of cefoxitin and imipenem on the emergence on multiresistant bacteria in the digestive flora

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient admitted to any medical or surgical department in the participating centre
* Documented urinary tract infection (other than cystitis), with or without bacteremia, caused by ESBL-producing E. coli susceptible in vitro to cefoxitin (minimal inhibition concentration <= 8 mg/L and /or diameter ≥ 19 mm according to CA-SFM 2015) and resistant to fluoroquinolones and to association trimethoprim-sulfamethoxazole. An E. Coli urinary tract infection is defined according to SPILF 2014 Clarification by a leucocytury ≥ 104/mL and clinical significant limit at 103 UFC/ml, for the men or the women.
* Medical examination prior to inclusion
* Informed consent signed by the patient
* Patient affiliated to a French Sécurité Social regimen

Exclusion Criteria:

* Serious infection (severe sepsis, septic shock)
* Pregnant or breast-feeding women
* Chronic kidney failure (creatinine clearance < 30 ml/min) and/or dialysis
* Hypersensibility to imipenem/cilastatine, to cefoxitine
* Hypersensibility to another antibiotics of cephalosporine class
* Hypersensibility to another antibiotics of carbapenem class
* Severe hypersensibility (ex :anaphylactic reaction, or serious cutaneous reaction) to all other antibiotics from beta lactamines family (ex : penicillins, monobactam)
* Treatment with ganciclovir and/or valproic acid
* Infection on the urinary cathether
* Empirical antibiotic therapy including an aminoglycoside
* Patient being treated with antibiotic(s) for another infection
* Patient participating to another interventional study
* Patient not compliant according to the investigator's opinion
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Control urine culture negative | 7 days after the end of treatment

SECONDARY OUTCOMES:
absence of fever | 3 days after the beginning of study treatment
  temperature lower than 38°C
presence of multiresistant bacteria in a rectal swab | 7 days after the end of treatment
Composite outcome measure consisting of resolution of clinical signs observed on diagnosis | 7 days after the end of treatment
  Absence of lower back pain, and/or absence of fictional burning, and/or absence of pollakiuria, and/or dysuria, and/or gross hematuria and/or abdominal pain

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France